CLINICAL TRIAL: NCT05297591
Title: Identifying Prognostic Variables for Persistent Upper Limb Dysfunctions After Breast Cancer Treatment: Longitudinal Cohort Study
Brief Title: Identifying Prognostic Variables for Persistent Upper Limb Dysfunctions After Breast Cancer Treatment
Acronym: UPLIFT-BC
Status: Recruiting | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, An De Groef, Prof. Dr, KU Leuven
Other Study IDs: s66248
Record Dates: First submitted 2022-03-17; First posted 2022-03-28 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: upper limb dysfunction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- breast cancer patients: Women and men diagnosed with breast cancer waiting for surgery
  Interventions: Other: assessment of UL function and prognostic factors

INTERVENTIONS:
Other: assessment of UL function and prognostic factors — clinical assessments and questionnaires

SUMMARY:
Breast cancer is the most frequently occurring cancer, assuming that it accounts for 29% of all new cancers in women (European Cancer Information System). The number of long-term survivors is increasing rapidly due to improving accuracy of the detecting methods, the early diagnosis and advances in cancer treatment.

The International Consortium for Health Outcomes Measurement Initiative described upper limb (UL) function as the health outcome that matters most for breast cancer survivors (BCS). 50% of BCS at 6 months post-radiotherapy suffer from of decreased UL function, i.e. difficulties in performing activities of daily living with the upper limb. Patients experiencing UL dysfunctions and other problems are less likely to be physically active. Given that physical inactivity is associated with an increased risk of mortality after breast cancer, taking away the barriers to physical activity (e.g. UL dysfunctions) is very important. Identifying these factors contributing to chronic UL dysfunction is important in terms of identifying targets for prospective evaluation and specific treatment approaches at specific time points during breast cancer treatment.

There is a need to rethink the follow-up strategy (besides the treatment of the cancer itself) and develop a clinical care pathway consisting of multifactorial screening instruments to identify women and men who are in need of extra rehabilitation efforts and specific rehabilitation goals to alleviate symptoms and side effects experienced by breast cancer survivors. This clinical care pathway should cover all aspects of the International Classification of Function, Disease and Health (ICF), a biopsychosocial framework that conceptualizes a person's level of functioning and bodily structures, activity and participation and contextual factors (including personal and environmental factors).

The present study aims to identify the factors, during and after breast cancer treatment, contributing to persistent Upper Limb (UL) dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery (mastectomy or breast conserving surgery; in combination with axillary lymph node dissection or sentinel node biopsy) for unilateral primary breast cancer or patients with oligometastatic breast cancer.
* Patients with a cognitive and language functioning enabling coherent Dutch communication between the examiner and the participant
* Patients who can comply with the protocol at baseline assessment and willing to provide written informed consent

Exclusion Criteria:

* BCS with widespread distance metastases, previous breast surgery, or planned bilateral surgery
* And/or with a diagnosis of a neurological or rheumatological condition,
* And/or BCS who are not available the entire duration of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from the population of breast cancer patients at the University Hospital Leuven
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Subjective upper limb function | Time frame up to 6 months post-radiotherapy
  quickDASH (0-100) questionnaire: An abbreviated version of the original DASH (Disabilities of the Arm, Shoulder and Hand) outcome measure. The questionnaire contains 11 items that measures an individual's ability to complete tasks, absorb forces and severity of symptoms, with a 5-point Linkert scale.
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Objective upper limb function | Time frame up to 6 months post-radiotherapy
  Accelerometry: duration of upper limb use (hours) during one week.
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of presence of skin deformities, asymmetry, presence of scapular winging or other scapular or shoulder deformities | Time frame up to 6 months post-radiotherapy
  Basic inspection of skin deformities, asymmetry, presence of scapular winging or other scapular or shoulder deformities.
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of pain intensity | Time frame up to 6 months post-radiotherapy
  Numeric Rating Scale (0-10) of pain intensity during movement during the week before assessment.
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of presence of neuropathic pain | Time frame up to 6 months post-radiotherapy
  Presence of neuropathic pain (yes/no):
  Douleur Neuropathique en 4 questions (DN4) is a questionnaire generated for identifying pain of predominantly neuropathic origin. The DN4 consists of 7 self-reporting questions and 3 clinical examinations. A scoring of ≥4/10 is considered as a positive result for neuropathic pain.
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of presence of sensory loss | Time frame up to 6 months post-radiotherapy
  Presence of sensory loss (yes/no) Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of presence of widespread pain | Time frame up to 6 months post-radiotherapy
  Presence of widespread pain (yes/no)
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of impact of pain on functioning | Time frame up to 6 months post-radiotherapy
  Brief Pain Inventory: the short version assesses the the impact of the pain on functioning.The Brief Pain Inventory is a valid multimodal scale for assessing pain in breast cancer patients.
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of Soft tissue stiffness index | Time frame up to 6 months post-radiotherapy
  The MyotonPRO assessment for soft-tissue stiffness and elasticity will take place at the pectoralis major, upper trapezius, infraspinatus and teres major region, from which a mean stiffness index (N/m) will be calculated.
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of Total relative arm volume (%) | Time frame up to 6 months post-radiotherapy
  Relative arm volume: Bilateral circumferential measurements using a perimeter will be performed.
  Water displacement method hand: Bilateral water displacement method using a volumeter filled with water and allowed to settle at room temperature will be performed.
  Afterwards the total volume (mL) can be calculated by taking the sum of the two measurements.
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of movement functions during a functional task | Time frame up to 6 months post-radiotherapy
  The 3D scapulothoracic and glenohumeral movements will be assessed using inertial sensors (MTw motion capture, Xsens Technologies, The Netherlands) at the endpoint (i.e. point of task achievement) of the performance of a functional task, the Upper Limb Function Test (ULIFT), which is a valid and reliable test to assess upper limb functionality in breast cancer patients.
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of Upper limb muscle strength (kg) | Time frame up to 6 months post-radiotherapy
  A hand-held dynamometer will be used to assess handgrip strength
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of Pain catastrophizing | Time frame up to 6 months post-radiotherapy
  Pain Catastrophizing Scale (0-52) : It is a self-report measure, consisting of 13 items scored from 0 to 4, resulting in a total possible score of 52. The higher the score, the more catastrophizing thoughts are present.
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of Self-efficacy | Time frame up to 6 months post-radiotherapy
  General Self-Efficacy Scale:This scale is a self-report measure of self-efficacy with 10 items (scored from 1-4). The total score is calculated by finding the sum of the all items. The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of Depression, Anxiety and Stress | Time frame up to 6 months post-radiotherapy
  Depression, Anxiety and Stress Scale (DASS-21) (range 0-132). The Depression, Anxiety and Stress Scale - 21 Items (DASS-21) is a set of three self-report scales designed to measure the emotional states of depression, anxiety and stress
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of Fear of movement | Time frame up to 6 months post-radiotherapy
  Adjusted 11-item Tampa Scale of Kinesiophobia. Items are scored from 1 (strongly disagree) to 4 (strongly agree). Thus, total scores range from 11-44 points with higher scores indicating greater fear of pain, movement, and injury
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of Body-perception | Time frame up to 6 months post-radiotherapy
  A self-developed Dutch version of the Fremantle Shoulder Awareness Questionnaire will be used.
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of Quality of Life | Time frame up to 6 months post-radiotherapy
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaires Core-30 item (EORTC QLQ-C30). The QLQ-C30 is a validated questionnaire that incorporates nine multi-item scales: five functional scales (physical, role, cognitive, emotional, and social); three symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of (Sub)optimal physical therapy care | Time frame up to 6 months post-radiotherapy
  Through a self-developed questionnaire, patients will be questioned whether they received no/suboptimal/optimal physical therapy care
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of treatment with Chemotherapy | Time frame up to 6 months post-radiotherapy
  no/taxanes/non-taxanes and neo-adjuvant/adjuvant (derived from the medical file) Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of treatment with Hormone therapy | Time frame up to 6 months post-radiotherapy
  no/aromatase inhibitor/no-aromatase inhibitor (derived from the medical file)
  Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.
Prognostic value of soft tissue adhesions | Time frame up to 6 months post-radiotherapy
  The 'Myofascial Adhesions in Patients after Breast Cancer (MAP-BC)'-tool will be used to assess the severity of soft tissue adhesions at the upper limb region (0-63) Assessment at pre-surgery baseline, 1 month post-surgery, 2 weeks post-chemotherapy (if applicable), 1 month post-radiotherapy and 6 months post-radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: An De Groef, Prof. Dr., Principal Investigator — KU Leuven
Locations (1):
- Universitair Ziekenhuis Leuven, Leuven, Belgium

REFERENCES:
- [Background] Hidding JT, Beurskens CH, van der Wees PJ, van Laarhoven HW, Nijhuis-van der Sanden MW. Treatment related impairments in arm and shoulder in patients with breast cancer: a systematic review. PLoS One. 2014 May 9;9(5):e96748. doi: 10.1371/journal.pone.0096748. eCollection 2014. PMID 24816774
- [Background] Berry DA, Cronin KA, Plevritis SK, Fryback DG, Clarke L, Zelen M, Mandelblatt JS, Yakovlev AY, Habbema JD, Feuer EJ; Cancer Intervention and Surveillance Modeling Network (CISNET) Collaborators. Effect of screening and adjuvant therapy on mortality from breast cancer. N Engl J Med. 2005 Oct 27;353(17):1784-92. doi: 10.1056/NEJMoa050518. PMID 16251534
- [Background] De Groef A, Meeus M, De Vrieze T, Vos L, Van Kampen M, Christiaens MR, Neven P, Geraerts I, Devoogdt N. Pain characteristics as important contributing factors to upper limb dysfunctions in breast cancer survivors at long term. Musculoskelet Sci Pract. 2017 Jun;29:52-59. doi: 10.1016/j.msksp.2017.03.005. Epub 2017 Mar 14. PMID 28319882
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] Ustun TB, Chatterji S, Bickenbach J, Kostanjsek N, Schneider M. The International Classification of Functioning, Disability and Health: a new tool for understanding disability and health. Disabil Rehabil. 2003 Jun 3-17;25(11-12):565-71. doi: 10.1080/0963828031000137063. PMID 12959329
- [Background] Yang EJ, Kim BR, Shin HI, Lim JY. Use of the international classification of functioning, disability and health as a functional assessment tool for breast cancer survivors. J Breast Cancer. 2012 Mar;15(1):43-50. doi: 10.4048/jbc.2012.15.1.43. Epub 2012 Mar 28. PMID 22493627
- [Derived] De Groef A, Vets N, Devoogdt N, Smeets A, Van Assche D, Emmerzaal J, Dams L, Verbeelen K, Fieuws S, Baets L. Prognostic factors for the development of upper limb dysfunctions after breast cancer: the UPLIFT-BC prospective longitudinal cohort study protocol. BMJ Open. 2024 May 15;14(5):e084882. doi: 10.1136/bmjopen-2024-084882. PMID 38754876